CLINICAL TRIAL: NCT06189612
Title: Is the Combination of Manual Therapy and Movement Control Exercises More Effective Than Manual Therapy and Standard Exercises in a Population of Patients With Chronic Neck Pain to Reduce Neck Disability? A Pilot Randomized Controlled Trial
Brief Title: Manual Therapy and Movement Control Exercises for Chronic Neck Pain. A Pilot Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hochschule Osnabruck (Other)
Collaborators: Medizinische Gesellschaft für Myofasziale Schmerzen e.V. (Unknown); Therapiecentrum Voxtrup - Praxis für Physiotherapie (Unknown); Facharztzentrum für Orthopädie, Unfallchirurgie und Rehabilitation des Bewegungssystems (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSOS/2023/9/15
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain; Temporomandibular Disorder
Keywords: Exercises; Motor control
MeSH Terms: conditions — Neck Pain; Temporomandibular Joint Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Three groups (msk + cervical motor control training, msk + orofacial motor control training, msk + standard exercises) will receive the protocol at the same time period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assessing clinician will be blinded to group allocation. Participants will be unaware of the hypothesis of this study to decrease performance biases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group1: Clinical reasoning-based physiotherapy + cervical movement control training (Experimental): Physiotherapeutic treatment is carried out based on the results of a subjective and physical examination performed at the outset. It may thus include various manual therapy treatment approaches targeting the maxillary and/or cervical or thoracic regions and adapted individually to each patient. In addition, one third of each treatment time is used to gradually teach patients the abnormal (positive) tests of the test battery for assessing motor control of the cervical region as a self-exercise for home use. To do this, patients are also given access via a quick response (QR) code to a website where they can find videos and instructions for the exact exercises that are in their home program.
  Interventions: Other: Clinical reasoning based physiotherapy + cervical movement control training
- Group 2: Clinical reasoning-based physiotherapy + orofacial movement control training (Experimental): Physiotherapeutic treatment is carried out based on the results of a subjective and physical examination performed at the outset. It may thus include various manual therapy treatment approaches targeting the maxillary and/or cervical or thoracic regions and adapted individually to each patient. In addition, one third of each treatment time is used to gradually teach patients the abnormal (positive) tests of the test battery for assessing motor control of the orofacial region as a self-exercise for home use. To do this, patients are also given access via a QR code to a website where they can find videos and instructions for the exact exercises that are in their home program.
  Interventions: Other: Clinical reasoning based physiotherapy + orofacial movement control training
- Group 3: Clinical reasoning-based physiotherapy + standard exercises (Active Comparator): Physiotherapeutic treatment is carried out based on the results of a subjective and physical examination performed at the outset. It may thus include various manual therapy treatment approaches targeting the maxillary and/or cervical or thoracic regions and adapted individually to each patient. In addition, one third of each treatment time is used to gradually teach patients general coordination- and strength exercises for the jaw and the cervical region as a self-exercise for home use. To do this, patients are also given access via a QR code to a website where they can find videos and instructions for the exact exercises that are in their home program.
  Interventions: Other: Clinical reasoning based physiotherapy + standard exercises

INTERVENTIONS:
Other: Clinical reasoning based physiotherapy + cervical movement control training — An individualized cervical motor control training based on the positive tests of the test battery introduced by Patroncini et al. (2014).
  Arms: Group1: Clinical reasoning-based physiotherapy + cervical movement control training
Other: Clinical reasoning based physiotherapy + orofacial movement control training — An individualized orofacial motor control training based on the positive tests of the test battery introduced by von Piekartz et al. (2017).
  Arms: Group 2: Clinical reasoning-based physiotherapy + orofacial movement control training
Other: Clinical reasoning based physiotherapy + standard exercises — A generalized training regimen based on exercises which are taught in physiotherapy training for the neck and scapula region preventing the overlap with exercises of the test batteries.
  Arms: Group 3: Clinical reasoning-based physiotherapy + standard exercises

SUMMARY:
Chronic neck pain is a common and highly prevalent clinical entity among the population. It causes a high economic and financial burden. Commonly people with neck pain present temporomandibular disorders (TMD). These conditions are closely correlated with each other. Several studies have shown that patients with neck pain do have abnormalities in motor control, endurance capacities, and strength of the cervical and orofacial area.

Several treatment modalities are available for neck pain that can be divided into pharmaceutical and non-pharmaceutical approaches. Among the non-pharmaceutical interventions, physiotherapy, manual therapy and exercises are of interest. The effect of treatment modalities is heterogeneous. Passive modalities often lack positive long-term outcomes.

Therefore, our trial aims to measure the effects of a combined treatment, consisting in manual therapy and a movement control training for the neck region or for the temporomandibular region, respectively. The implementation of the temporomandibular movement control training is based on the assumption that there might be crossover effects between both regions, i.e., convergence of cervical and trigeminal sensory afferents between these two regions.

We designed a parallel randomized controlled trial (RCT) with three intervention arms and a blinded assessor for outcomes that are clinician performed. This study is a pilot trial, so each group is expected to consist of 15 subjects. Both female and male patients between the ages of 18 and 65 will be included. Participants must suffer from idiopathic chronic neck pain (at least 3 months) and may also have symptomatic TMD disorders. The Primary Outcome will be neck pain disability measured by the Neck Disability Index (NDI). Secondary Outcomes will be Diagnostic Criteria (DC)/TMD (Axis I and Axis II), range of motion (CROM, FRT), CVA, PPT, CCFT, and both cervical and orofacial test batteries to assess motor control in each region.

Patients are randomly assigned to one of the three intervention groups using a computer-generated sequence which is concealed. The three groups are: 1) clinical reasoning (CR) based physical therapy + cervical motor control training, 2) CR based physical therapy + orofacial motor control training, 3) CR based physical therapy + general coordination and strengthening exercises for the jaw and neck region.

Prior to the start of treatment, participants will undergo an eligibility assessment. If the participant meet the inclusion criteria, the baseline assessment is conducted, and the treatment is planned following the prescription for physiotherapy in Germany. Treatment will comprise six 30-minute treatment sessions, which take place once a week over a period of 6 weeks. Upon completion of the six treatment sessions, the final examination is conducted, which includes the same assessments as the initial examination.

DETAILED DESCRIPTION:
Considered from an epidemiologic perspective, musculoskeletal (MSK) disorders are highly burdensome and one of the most leading causes for illness especially in work life. Especially low back pain and neck pain are highly prevalent, even ranging among the top ten of health issues worldwide. Patients with neck pain (NP) often present headaches and orofacial pain (OFP) (including temporomandibular disorders). Most of these disorders can occur concomitantly and overlap to a greater extent. Therefore NP, headache and OFP are generally investigated together.

Since the causes for neck pain are multicausal, several treatment approaches exist, which can be divided into pharmaceutical and non-pharmaceutical modalities. The non-pharmaceutical approaches are further divided into surgical and non-surgical. However, in clinical practice, these different approaches are often combined.

In the domain of musculoskeletal therapy, the treatment modalities for chronic neck pain range from passive approaches, for example spinal manipulation (SMT) or myofascial trigger point therapy, to biopsychosocial approaches like pain neuroscience education (NPE). Exercise therapy is another treatment modality with good effect for this condition. Exercise therapy can further be divided into strength training, endurance training and coordination training. Motor control training (MCT) is an important treatment option.

However, clinical trials often analyze single approaches (stand-alone-modalities), while in clinical practice these approaches are frequently combined. Therefore, our trial aims to analyze the effects of manual therapy combined with a motor control training program. Our trial will respond several clinical/research questions.

Q1) Does the combination of clinical reasoning-based manual therapy and movement control for the neck region (G1) or the orofacial region (G2), respectively, generate additional effects in terms of lowering the NDI score (main outcome) and improving CROM, FRT, CVA, PPT and CCFT (secondary outcomes) compared to manual therapy and standard exercises (usual care) (G3)?

Q2) Are the summary scores of the orofacial test battery and the neck test battery significantly improved (which means lower scores) in the groups that received the targeted interventions (G1 and G2) compared to the group (G3)?

Q3) Is there an association between the neck and orofacial test battery performances (scores)?

The aim of the present pilot randomized controlled trial is to determine the potential additional benefits of movement control exercises added to usual care. Therefore, movement control exercises are anticipated to be more effective than standard exercises.

Sample size: Since there are no comparable trials, there are no known effect sizes of the interventions of interest to provide an accurate sample size calculation. Therefore, this present project will provide evidence of this effect for future studies and will be set up as a pilot trial. For this reason, we set a sample size of n = 15 per group, as recommended by the literature regarding sample sizes for pilot trials.

Procedure. The patients will be recruited by an orthopaedic physician in a clinical practice. A trained physiotherapeutic assessor will determine subjects' eligibility and perform the assessments at the baseline and after the treatments. Demographic data will be collected. Additionally, the primary outcome, neck disability measured with the Neck Disability Index (NDI) will be assessed. The secondary outcomes include the tests and outcomes measures provided by the DC/TMD (Axis I and Axis II), neck range of motion (CROM), Flexion rotation test (FRT), Craniovertebral Angle (CVA), Pressure Pain Thresholds (PPT), Craniocervical flexion test (CCFT), and both cervical and orofacial test batteries to assess motor control in each region which are videotaped. After baseline assessments, randomization will take place and treatments will start. Treatment will comprise six 30-minute treatment sessions, which take place once a week over a period of 6 weeks. After the last session of treatment, measurements will be again conducted.

Randomization. A randomization sequence stratified by age (18-30, young adult; 31-45, adult; 46-60, older adult) and gender (female and male) was generated by a computer software by a third party not involved in subjects' recruitment or treatment. This sequence was placed in opaque, sealed and numbered envelopes to warranty concealment from the research team. When is ensured that the patient is eligible, the therapist will open the envelope that contains the sequence to indicate the group assignment

Treatments. The patients will receive six treatments. Based on the analysis of the movement control tests, a link will be sent to the patients to unlock videos containing the movement tests that were assessed as having poor performance (positive tests), so the patient can train those specific movements. The movement tests that will be given to each patient will depend on the group assignment. The videos are similar to the movement control tests for training purposes. The description of the treatments will be described in section treatments

Timeline. After the baseline examination, patients receive six treatments, according to the doctor's prescription. These are scheduled once or twice a week. After the sixth treatment, the post-interventional final examination will be performed approximately 4-8 weeks after the pre-interventional assessment. Thus, the timeline respects the medical prescription according to German statutory health insurance conditions.

Compliance and contamination. At the beginning of every treatment session, the therapist will ask the patients how many times they trained to protocolize compliance with the treatment.

Positive and negative consequences for the test subjects: Since the exercises are designed to improve movement control, there are no high loads to expect and therefore, the risk for the patients is minimal. Manual therapy is based on clinical reasoning, respecting potential irritability and severity, and therefore reduces the risk of adverse treatment reactions. However, if adverse effects occur, the physicians who sent the patients will be consulted, and if it is possible, an appointment will be scheduled quickly.

Statistical analysis . To determine whether the combination of clinical reasoning-based manual therapy and movement control training programs for the neck region (G1) or the orofacial region (G2), generate additional effects in terms of lowering the NDI score (main outcome) and improving CROM, FRT, CVA, PPT and CCFT (secondary outcomes) compared to manual therapy and standard exercises (G3)(Q1), we will compute mean change scores (second assessment minus baseline) and will perform an Analysis of Variance (ANOVA) to reveal whether statistically significant differences between groups might exist. Bonferroni Post-hoc test (or Games Howell) will complement the omnibus ANOVA in order to determine where the differences between groups exist. Normal distribution will be tested by using Kolmogorov Smirnov test and homogeneity of variance will be tested with Levene's test.

If the assumptions of ANOVA are not met, we would run a non-parametric equivalent model using Kruskal-Wallis-test or Robust ANOVA to determine our p-values. We hypothesize that the NDI's mean score will be significantly lower in the interventional groups performing movement control programs (G1, G2) compared to G3 which receives usual care (manual therapy and standard exercises). We further expect the secondary outcomes (detailed description in the section outcome measures) to be significantly improved in G1 and G2 compared to G3. All primary and secondary outcomes will be considered as continuous variables for analyses.

Q2) Are the summary scores of the orofacial test battery and the neck test battery significantly improved (which means lower scores) in the groups that received the targeted interventions (G1 and G2) compared to the group (G3)?

Since the movement control groups (G1 and G2) will receive a training program that is guided by the positive scored tests in the neck test battery (G1) or the orofacial test battery (G2), we expect the scores of these test batteries to be significantly improved after the intervention compared to the control group that receives standard care. In statistical terms, we expect the scores to be significantly lower in G1 and G2. For this purpose, the total scores of the test batteries will be calculated by adding up the positive tests. For the cervical tests, that means a range from 0 to 13 and for the orofacial battery a range from 0 - 8, respectively. As the number of positive tests is added together for the total score, this variable can be regarded as discrete. Single Poisson regression analyses will be used to determine differences between groups on the summary scores of the orofacial test battery and the neck test battery. The dependent variables are the summary scores and the independent variables would be the groups.

The alpha level will be set to p=0.05 for all analyses.

Q3) Is there an association between the neck and orofacial test battery performances (scores)? The summary scores of the test batteries (ranging from 0-13 for the cervical test battery and from 0-8 for the orofacial test battery) will be used for a regression model. In statistical terms, we wonder if it possible to predict the neck summary score (dependent variable) by knowing the orofacial test summary score (independent variable) by other covariables of interest (age, gender, pain chronicity). Therefore, the assumptions of a Poisson regression will be considered.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 - 65 years of age
* being diagnosed with idiopathic chronic neck pain (>= 3 month)
* scoring minimum >= 15 in the NDI
* linguistic (german) and cognitive ability to fully understand the questionnaires and exercise instructions.

Exclusion Criteria:

* presence of neurological symptoms of the upper limb
* presence of elapsed fractures or surgeries in the past half year in the head, jaw or cervical region
* medical interventions in these regions
* systemic inflammatory conditions requiring systemic-acting drugs
* Central Sensitization Index (CSI) score > 40 points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | baseline, final evaluation (6 treatments (6-8 weeks) after the baseline measurement)
  This is a 10-item self-report questionnaire designed to assess the extent to which neck pain interferes with activities daily living. The Neck Disability Index is a validated, reliable and responsive tool. The score ranges from 0 and 50 points, the achieved value is divided by the maximum score of 50 and multiplied by 100. This is how the score of the NDI is calculated. A higher value equals higher disability.

SECONDARY OUTCOMES:
Diagnostic criteria for temporomandibular disorders DC/TMD (Axis I and Axis II) | baseline, final evaluation (6 treatments (6-8 weeks) after the baseline measurement)
  Axis I: In addition to the "TMD Pain Screener" and the "Symptom Questionnaire", the physical examination is carried out according to a standardized protocol (Schiffmann et al. 2014). Symptoms are localized and then the position of the anterior teeth and the opening pattern are assessed. In the measurement of the range of motion, the mouth opening, laterotrusion to the left and right and protrusion are taken into account. In addition to the range of motion in mm, it is also assessed whether any (known) pain has occurred. Next, joint noises are assessed during the jaw movements. In addition, it is assessed whether a blockage occurs during the examination.
  Axis II: Axis II is used to identify psychosocial characteristics. The following questionnaires are used for this purpose: Graded chronic pain scale (v2), Jaw Functional Limitation Scale-8 (JFLS-8), JFLS-20, Patient Health Questionnaire-4 (PHQ-4), PHQ-9, Generalized Anxiety Disorder Scale-7 (GAD-7), PHQ-15, Oral Behaviors Checklist.
Craniovertebral angle | Time Frame: baseline, final evaluation (6 treatments (6-8 weeks) after the baseline measurement)
  In order to measure the craniovertebral angle a picture of the patient sitting in his habitual position is taken from the side. The camera position is standardized, thus the angle and the distance to the patient is always the same. To determine the craniovertebral angle a horizontal line is drawn through the spinous process of C7. A second line connects the tragus of the ear and C7. The angle formed by these two lines is measured using a digital imaging software. The smaller the angle, the stronger the forward head posture.
Pressure Pain Threshold | baseline, final evaluation (6 treatments (6-8 weeks) after the baseline measurement)
  Pressure pain sensitivity will be evaluated by assessing the pressure pain threshold (PPT). This is the minimum amount of pressure that induces pain or a feeling of discomfort. The PPT will be measured within several masticatory muscles and neck muscles using the NOD device with the algometry function. The value is measured in kilopascals (kPa) and a higher value means a better result.
Craniocervical flexion test | baseline, final evaluation (6 treatments (6-8 weeks) after the baseline measurement)
  The deep cervical flexor muscles are assessed performing a modified craniocervical flexion test (CCFT) via the Nod-device. The patient will lay supine with the neck positioned on the Nod-device and the connected magnetic pad. The patient will then be instructed to perform a gentle and slow movement, like a "yes" head-nodding action. The test consists of two steps. During step one, the maximum force of the head-nodding action will be measured in Newton (N). In the second step the patient is asked to hold the nod-movement for 10 seconds at 20%, 40%, 60%, 80% and 100% of the maximal force . There is a range of 10% above or below the target value, which is also considered correct. The NOD-Device is used to determine the percentage of time in which the power of the head-nodding movement is in the target range and thus a higher score equals a better performance of the deep cervical flexor muscles.
Cervical test battery to assess movement control in the cervical region | baseline, final evaluation ( (6 treatments (6-8 weeks) after the baseline measurement)
  The 13 tests to assess motor control of the cervical region are carried out as described by Patroncini et al. (2014). The assessment is based on the video recordings of the test performance. Each test is assessed as either correct or incorrect. The criteria for judging a test as correct or incorrect are defined in advance according to the guidelines provided by Patroncini et al. 2014. Therefore, a standardized videotaping set-up is installed in a room in which every measurement will take place. After the baseline assessment, the therapist will assess the videotaped tests considering the strictly defined conditions provided by Patroncini et al. 2014.
Orofacial test battery to assess movement control in the orofacial region | baseline, final evaluation ( (6 treatments (6-8 weeks) after the baseline measurement)
  The eight tests to assess motor control of the orofacial region are carried out as described by Piekartz et al. (2017). The assessment is based on the video recordings of the test performance. Each test is scored from 1 to 6 according to the occurrence of associated movements or the incomplete execution of the movement. Like above, the videotaping is standardized like in the trial of Piekartz et al. (2017). Videotaping of motor control is a reliable technique (Franki et al. 2015).
Upper and global cervical range of motion | baseline, final evaluation (6 treatments (6-8 weeks) after the baseline measurement)
  - Upper neck range of motion (ROM) will be measured by carrying out the Flexion Rotation Test (FRT) to the left and right side. Additionally, the global movements of the cervical spine will be measured: flexion, extension, lateral-flexion and rotation. All measurements will be performed using a "Neck Care" device, thus the ROM is measured in degrees. The higher the value, the larger the ROM of the cervical spine.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Armijo-Olivo, PhD, Principal Investigator — Hochschule Osnabruck
Locations (1):
- Hochschule Osnabrück, Osnabrück, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patroncini M, Hannig S, Meichtry A, Luomajoki H. Reliability of movement control tests on the cervical spine. BMC Musculoskelet Disord. 2014 Nov 29;15:402. doi: 10.1186/1471-2474-15-402. PMID 25432070
- [Background] von Piekartz H, Stotz E, Both A, Bahn G, Armijo-Olivo S, Ballenberger N. Psychometric evaluation of a motor control test battery of the craniofacial region. J Oral Rehabil. 2017 Dec;44(12):964-973. doi: 10.1111/joor.12574. Epub 2017 Sep 30. PMID 28892191
- [Background] Franki I, Van den Broeck C, De Cat J, Molenaers G, Vanderstraeten G, Desloovere K. A study of whether video scoring is a reliable option for blinded scoring of the Gross Motor Function Measure-88. Clin Rehabil. 2015 Aug;29(8):809-15. doi: 10.1177/0269215514558642. Epub 2014 Nov 21. PMID 25416132